CLINICAL TRIAL: NCT06112834
Title: Tolerability and Immunogenicity of a Single 40-µg Dose of Recombinant Botulinum Vaccine A/B (rBV A/B) for the Production of BabyBIG® in Volunteers With Existing Botulinum Immunity
Brief Title: Tolerability and Immunogenicity of a Single 40-ug Dose of rBV A/B for the Production of BabyBIG®
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: California Department of Public Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: rBV A/B-CL-003
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Botulism
MeSH Terms: conditions — Botulism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vaccine (Experimental): rBV A/B
  Interventions: Biological: rBV A/B

INTERVENTIONS:
Biological: rBV A/B — Recombinant Botulinum Vaccine A/B, rBV A/B

SUMMARY:
This Phase 2, open-label, uncontrolled study designed to evaluate safety, tolerability, and immunogenicity of a single dose of rBV A/B in healthy participants previously immunized with pentavalent botulinum toxoid (or pentavalent botulinum toxoid and rBV A/B) for occupational protection will be conducted to collect source plasma for potential use in the production of BabyBIG and to evaluate safety and immunogenicity of the vaccine in these participants over a 12-week period, with a follow-up safety assessment at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Have received pentavalent botulinum toxoid (or pentavalent botulinum toxoid and rBV A/B) for occupational protection under BB IND 0161 (or BB-IND-0161 and IND 015155)
2. Are 18 to 69 years old at the time of consent
3. Are healthy and have an acceptable medical history (defined as individuals who are free from significant cardiac, pulmonary, gastrointestinal, hepatic, renal, hematological, neurological, infective, muscular, infectious, rheumatic, immunological, or psychiatric diseases, as determined at screening) that will not interfere with the objectives of the study
4. Meet the participant suitability requirements and recommendations for source plasma donors
5. Participants of childbearing potential:

   * Must have negative pregnancy test at screening and within 24 hours prior to vaccination.
   * Must agree to not become pregnant until after the last plasma donation or until after the Week 12 visit (whichever occurs last).
   * Must agree to use at least one form of highly effective birth control starting 30 days prior to rBV A/B administration through the end of the study. Acceptable forms of contraception include intrauterine device, birth control pills, injectable birth control, implantable birth control device, or any other U.S. FDA approved contraceptive method or a monogamous relationship with partner who has been vasectomized for at least 6 months prior to participant's enrollment or sexual abstinence.
6. To be considered of non-childbearing potential, participants must be menopausal (no menstrual period for at least 12 months prior to screening) or be surgically sterile
7. Are able to understand the requirements of the study, have provided written informed consent as evidenced by signature on an informed consent form (ICF) approved by the appropriate Institutional Review Board (IRB), and have agreed to abide by the study restrictions and return for the required assessments
8. Agree to complete the participant home diary on a daily basis for 7 days post vaccination, as well as to report any severe adverse events (AEs) and serious AEs (SAEs), including serious new onset chronic illnesses (NOCIs) and concomitant medications during the study period
9. Have provided written authorization for use and disclosure of protected health information
10. Agree not to donate blood or blood products (outside of study procedures) until after the last plasma donation or until the Week 12 visit (whichever occurs last)
11. Have personal health insurance

Exclusion Criteria:

1. Are pregnant or nursing
2. Have a history of laboratory evidence of syphilis, acquired immunodeficiency syndrome, Creutzfeldt-Jakob disease, or infection with human immunodeficiency viruses (HIV) 1 or 2, human T-cell lymphotropic virus 1, hepatitis B virus (HBV), or hepatitis C virus (HCV)
3. Have had a prior severe (Grade 3 or higher) local or severe (Grade 3 or higher) systemic reaction to last immunization with PBT
4. Have had a prior severe immediate hypersensitivity reaction or severe systemic reaction on Day 0 to last vaccination with rBV A/B
5. Have known allergy to aluminum, yeast, or other components of the vaccine
6. Have donated one or more units of blood or undergone plasmapheresis within 49 days prior to enrollment
7. Have received a blood product or immunoglobulin within 6 months prior to enrollment or plans to receive such products during the study period (exclusive of returned red blood cells as part of the plasmapheresis procedure). For participants who choose to donate plasma, this will apply until their last plasma donation or at the Week 12 visit (whichever occurs last)
8. Have received licensed nonliving vaccine within 14 days prior to enrollment, or licensed live vaccine within 60 days prior to enrollment
9. Have received nonliving vaccine authorized for emergency use only within 14 days prior to enrollment, or living vaccine authorized for emergency use only within 60 days prior to enrollment
10. Have received investigational products (drugs, biologics, vaccines [except for those authorized for emergency use only per exclusion criterion 9], or implantable devices) within 60 days prior to enrollment or plans to receive experimental products at any time during the study period. For participants who choose to donate plasma, this will apply until their last plasma donation or at the Week 12 visit (whichever occurs last)
11. Have received prescription immunosuppressive or immunomodulatory agents, including parenteral, inhaled, or oral corticosteroids within 3 months of enrollment or plans on receiving such therapy at any time during the study period. For participants who choose to donate plasma, this will apply until their last plasma donation or at the Week 12 visit (whichever occurs last), with the exceptions mentioned below:

    * Participants who have used prescription topical steroids may be enrolled 2 weeks after the therapy is completed
    * Intra-articular, bursal, or tendon injectable steroids are permitted
    * Any over-the-counter topical steroid use is permitted
    * Ophthalmic and intranasal steroids are permitted
12. Have received cytotoxic therapy at any time in the previous 5 years before enrollment
13. Have an active systemic or recurrent disease that would place the participant at unacceptable risk of injury, require hospitalization, or require surgical intervention (This includes active mental illness or history of mental illness not responsive to treatment.)
14. Have a history of alcohol or drug abuse or dependence within 12 months of enrollment
15. Have past, present, or suspected illicit injection drug use
16. Have inflammatory, vasculitic, or rheumatic disease, including systemic lupus erythematosus, polymyalgia rheumatica, rheumatoid arthritis, or scleroderma (Stable osteoarthritis treated with physical therapy and nonsteroidal anti-inflammatory drugs is not an exclusion criterion.)
17. Have any acute or chronic neuromuscular or neurologic disorder
18. Have clinically confirmed hepatic or renal insufficiency
19. Have uncontrolled hypertension, as defined a systolic blood pressure greater than 160 mmHg and diastolic blood pressure greater than 90 mmHg
20. Have moderate to severe asthma, chronic obstructive pulmonary disease, or other significant pulmonary disease
21. Have a seizure disorder
22. Have moderate or severe illness or oral temperature of 100.4°F or greater within 3 days prior to enrollment
23. Have any positive result for SARS-CoV-2 (COVID-19) using an FDA-cleared or FDA-authorized test within 14 days of enrollment
24. Be unsuitable for participation in this study for any reason, as assessed by the investigator

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-07-09 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
Proportion of Subjects Achieving Equal to or Greater Than 4-Fold Increase in Neutralizing Antibody Concentration (NAC) | Week 0 to Week 4
  The primary immunogenicity endpoint is the proportion of participants achieving a four times or greater increase in NAC by Week 4 compared with Week 0. A positive response will be defined as achieving this level of increase in at least 50% of the participants for botulinum toxin type A and type B.

SECONDARY OUTCOMES:
Proportion of Subjects Achieving 2-Fold Increase in Area Under the Plasma Concentration-Time Curve in Neutralizing Antibody Concentration (NAC) | Week 0 to Week 12
  The proportion of participants achieving two times increase in the area under the plasma concentration-time curve between Week 0 and Week 12 in NAC in comparison to a straight-line extension of the Week 0 NAC to Week 12. A positive response will be defined as achieving this level of increase in at least 50% of participants for botulinum toxin type A and type B.
Proportion of Subjects Achieving Equal to or Greater Than 3-Fold Increase in Neutralizing Antibody Concentration (NAC) | Week 0 to Week 4
  The proportion of participants achieving a three times or greater increase in NAC by Week 4 compared with Week 0. A positive response will be defined as achieving this level of increase in at least 50% of the participants for botulinum toxin type A and type B.

OTHER OUTCOMES:
Volume of Plasma Collected with Anti-Botulinum Toxin Type A and Anti-Botulinum Toxin Type B Antibody Titers | Week 0 to Week 12
  The volume of source plasma containing neutralizing antibodies against botulinum toxin type A and type B collected by plasmapheresis for use in BabyBIG manufacture.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - California Department of Public Health, Richmond, California
  - Battelle Biomedical Research Center, West Jefferson, Ohio

IPD SHARING:
Plan to Share IPD: No